CLINICAL TRIAL: NCT03551249
Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier Disruption for the Treatment of High Grade Glioma in Patients Undergoing Standard Chemotherapy
Brief Title: Assessment of Safety and Feasibility of ExAblate Blood-Brain Barrier (BBB) Disruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BT008
Record Dates: First submitted 2018-04-17; First posted 2018-06-11 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Focused Ultrasound (FUS) (Experimental): The ExAblate Model 4000 Type 2 system is intended for use as a tool to induce localized and temporary blood-brain barrier disruption in patients with glioblastoma undergoing initial standard of care chemotherapy.
  Interventions: Device: Focused ultrasound (FUS)

INTERVENTIONS:
Device: Focused ultrasound (FUS) — FUS involves the application of acoustic energy at low frequencies from over 1000 individual transducers into distinct body targets.
  Other Names: ExAblate, Type 2

SUMMARY:
The purpose of this study is to evaluate the safety of the ExAblate Model 4000 Type 2 used as a tool to disrupt the BBB (blood brain barrier) in patients with high grade glioma undergoing standard of care therapy.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-arm study to establish the safety and feasibility of BBB (blood brain barrier) disruption along the periphery of tumor resection cavity using the ExAblate Neuro Model 4000 Type 2 (220 kHz) system. For this study, patients will be eligible to enroll in the study prior to beginning the planned adjuvant TMZ chemotherapy phase of treatment. Of note, only patients who are deemed eligible for adjuvant TMZ will be eligible for enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is eligible for adjuvant temozolomide (TMZ) treatment based on the current standard of care.
2. Men or women age between 18 and 80 years, inclusive.
3. Able and willing to give informed consent.
4. Grade IV glioma (GBM)
5. Combined radiation/TMZ treatment is completed based on the prescribed standard of care regimen.
6. Karnofsky rating 70-100.
7. Able to communicate during the ExAblate BBBD (Blood Brain Barrier Disruption) procedure.
8. Able to attend all study visits (i.e., life expectancy of at least 3 months).

Exclusion Criteria:

1. Patients presenting with the following imaging characteristics:

   i. Evidence of acute intracranial hemorrhage.
2. The sonication pathway to the tumor involves:

   i. Extensive scalp sores. ii. Clips or other metallic implanted objects in the skull or the brain (brain implants)
3. The subject presents with symptoms and signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, and papilledema).
4. Patients with cerebellar or brainstem tumors.
5. Patients with positive HIV status.
6. Significant depression not adequately controlled with medication and at potential risk of suicide.
7. Patient receiving bevacizumab (Avastin) therapy.
8. Patients receiving treatment with corticosteroid doses greater than dexamethasone 24 mg daily (or equivalent).
9. Patients undergoing other concurrent therapies such as chemotherapy wafers, immunotoxins delivered by convection-enhanced delivery, regionally administered gene and viral therapies, immunotherapies, focal irradiation with brachytherapy, stereotactic radiosurgery, laser interstitial thermotherapy, and tumor treatment fields therapy.
10. Cardiac disease or unstable hemodynamics including:

    i. Documented myocardial infarction within six months of enrollment. ii. Unstable angina on medication. iii. Congestive heart failure. iv. Left ventricular ejection fraction <50%. v. History of a hemodynamically unstable cardiac arrhythmia. vi. Cardiac pacemaker.
11. Severe hypertension (diastolic BP > 100 on medication).
12. Anti-coagulant therapy, or medications known to increase risk of hemorrhage within washout period prior to treatment.
13. History of a bleeding disorder, coagulopathy or with a history of spontaneous tumor hemorrhage.
14. Cerebral or systemic vasculopathy, including intracranial thrombosis, vascular malformation, cerebral aneurysm or vasculitis.
15. History of drug or alcohol use disorder.
16. Active seizure disorder or epilepsy (seizures despite medical treatment).
17. Known sensitivity to gadolinium-based contrast agents.
18. Known sensitivity to DEFINITY® ultrasound contrast agent or perflutren.
19. Contraindications to MRI such as non-MRI-compatible implanted devices.
20. Large subjects not fitting comfortably into the MRI scanner.
21. Difficulty lying supine and still for up to 4 hours in the MRI unit or claustrophobia.
22. Positive pregnancy test (women of childbearing potential).
23. Severely impaired renal function or on dialysis.
24. Cardiac shunt.
25. Subjects with evidence of cranial or systemic infection.
26. Subjects with significant liver dysfunction, e.g., history of cirrhosis or active hepatitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Device and procedure related adverse events | Throughout the study, approximately 12 months.
  The number and severity of device and BBB disruption procedure related adverse events will be evaluated and classified according to the CTCAE

SECONDARY OUTCOMES:
Feasibility of repeated BBB disruption will be evaluated through assessment of post-procedure contrast-enhanced magnetic resonance (MR) imaging | At the time of each ExAblate MRgFUS procedure
  The repeatability of BBB disruption will be evaluated at each of the 6 procedures and will be evaluated through assessment of post-procedure contrast-enhanced MR imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Woodworth, MD, Principal Investigator — University of Maryland
Locations (4):
- United States (4):
  - University of Maryland, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woodworth GF, Anastasiadis P, Ozair A, Chabros J, Bettegowda C, Chen C, Gerstl JVE, Douville C, Mekary RA, Smith TR, Meng Y, Hawkins C, Pople CB, Abrahao A, Llinas M, Heyn C, Bunevicius A, Rezai AR, Ball AJS, Henry K, Sahgal A, Torio E, Ren H, Ahmad H, Arora H, Eisenberg H, Perry J, Carpenter JS, Hynynen K, Pham LC, Anketell MB, Lim-Fat MJ, Xu Z, Cifarelli CP, Sheehan JP, McDannold NJ, Gandhi D, Golby AJ, Lipsman N. Microbubble-enhanced transcranial focused ultrasound with temozolomide for patients with high-grade glioma (BT008NA): a multicentre, open-label, phase 1/2 trial. Lancet Oncol. 2025 Dec;26(12):1651-1664. doi: 10.1016/S1470-2045(25)00492-9. PMID 41308679